CLINICAL TRIAL: NCT05853809
Title: Clinical Effect of FeNO Measurement for Asthma Treatment in Primary Care: A Real-world Cluster-randomised Controlled Trial
Brief Title: Cluster-Randomized Asthma FeNO Trial
Acronym: CRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Region Stockholm (Other Government)
Collaborators: Uppsala University (Other); Karolinska Institutet (Other); Universidade do Porto (Other); Niox Group Plc (Unknown)
Responsible Party: Principal Investigator, Jörgen Syk, Director of Postgraduate Studies, Intern and Resident Physicians, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00919
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Exhaled nitric oxide; FeNO; Exacerbations; Asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FeNO measurement (Active Comparator): Anti inflammatory treatment guided by measurement of airway inflammation (FeNO).
  Interventions: Diagnostic Test: FeNO measurement
- Usual care (No Intervention)

INTERVENTIONS:
Diagnostic Test: FeNO measurement — FeNO measurement to guide anti-inflammatory asthma treatment
  Arms: FeNO measurement

SUMMARY:
Asthma is a chronic inflammatory respiratory disease that affects people of all ages and of both sexes. It is a common disease and is present in 8-10 % of the population. Despite drug treatment, many patients have poor control of their asthma with an impact on quality of life and restriction of daily activities. The purpose of this study in primary care is to investigate if measurement of airway inflammation (FeNO) can improve the treatment results and the overall care of adult patients with asthma. The main question in the study is whether the use of FeNO measurements can reduce the number of deterioration periods. The study is conducted under real clinical conditions where the effect of the intervention is measured (pragmatic intervention study). Eight to twelve primary health care centers with functional asthma / COPD clinics are selected within the Stockholm County and are randomly assigned to two groups with four to six primary health care centers each, an active group and a control group (cluster randomization). Instruments for FeNO measurements are made available to the active group and this group is also trained on FeNO measurements and how the value should be interpreted and used to control the treatment, while the control group continues to take care of their asthma patients as usual. The study can lead to improved treatment decisions and patients gaining an increased understanding of their asthma by being informed on the actual degree of inflammation in the airways. Optimized treatment can provide better asthma control with increased quality of life and fewer periods of deterioration, which results in reduced burden on healthcare and lower costs for patients and society.

DETAILED DESCRIPTION:
Cluster-Randomized Asthma FeNO Trial (CRAFT)

Clinical effect of FeNO measurement for asthma treatment in primary care: A real-world cluster-randomised controlled trial

Jörgen Syk, Hanna Sandelowsky, Björn Stridh, Kjell Alving

Overview of the field

The prevalence of asthma has increased in the last decades and seems to be increasing among children in Sweden also in the 21st century. A study performed by the Institute of Environmental Medicine at the Karolinska Institute, in collaboration with the National Board of Health and Welfare, showed that the prevalence of physician-diagnosed asthma increased between the years 2003 and 2011: from 6.1% to 9.5% among four-year-olds and from 6.4% to 8.9% among twelve-year-olds [1]. This likely portends a continued increase of the asthma prevalence among the adult population as well. The reason for the increase of allergy and asthma is likely to be multifactorial and therefore difficult to counteract at a societal level. Instead, healthcare must be developed to effectively diagnose and treat the increasing number of patients.

In the early 2000s, major hope was placed in combination inhalers (corticosteroid + long-acting beta-2 agonist) within asthma care, and prescription of these increased dramatically. However, studies have shown that the proportion of patients with controlled asthma has not increased after the introduction of such inhalers [2, 3], while the costs for asthma medication have increased drastically instead. Within the last ten years, the need has been identified for better characterisation of patients with asthma symptoms, as the asthma disease is heterogeneous and also varies over time. Particular interest has been raised in biomarkers like the fraction of exhaled nitric oxide, FeNO, and blood eosinophil levels (B-Eos) [4-6].

Currently, FeNO is the most commonly used clinical biomarker of asthma, although the method is not established within Swedish primary care. However, the British authority NICE (National Institute of Health and Care Excellence) states, in its 2017 guidelines on asthma, that FeNO should be used in asthma diagnosing and in treatment follow-up for patients with remaining symptoms despite treatment with inhaled corticosteroids (ICS) [7]. FeNO is a marker of type-2 inflammation in the airways, more specifically of mechanisms induced by interleukin (IL)-4 and IL-13. Dupilumab, a biological drug blocking the effect of IL-4/IL-13, has recently been approved within the EU as add-on maintenance treatment in severe asthma, but only for patients with detectable persistent type-2 inflammation, i.e., elevated FeNO and/or B-Eos.

FeNO, unlike B-Eos, correlates strongly with the degree of hyperreactivity to methacholine and mannitol [8], and elevated FeNO is a reliable predictor of clinical response to use of ICS [9]. FeNO usually decreases with use of ICS, except in cases of high allergen exposure [10, 11]. The FeNO value may thus be a very good starting point in the dialogue between a physician and a patient regarding treatment adherence and environmental aspects, such as exposure to furred pets.

Preliminary results

Our application is preceded by many years' research activity within the field by the group. We began with a pilot study at a primary healthcare centre to test a treatment algorithm guided by FeNO values. We could show that FeNO drops to normal levels following increased use of ICS, so long as allergen exposure is not too high [11].

Strengthened by these results, we moved on to a multi-centre study (NOAK) within primary care, with the Stockholm County Council as the main financier [12]. In this study, 187 adult patients with allergic asthma were randomised to an active group (FeNO-guided treatment) or a control group (usual care, mainly guideline-based) at 17 healthcare centres in central and southern Sweden. The patients were followed for 12 months, with 5 visits to their healthcare centre. The treatment was stepped up in the same way in both groups and included ICS and anti-leukotrienes. In this study, we could show a significantly larger improvement of asthma control (Juniper Asthma Control Questionnaire) and a decrease in the number of moderately severe exacerbations in the FeNO-guided group as compared with the control group, without any increase in average drug use. Internationally, several similar studies have been performed, and meta-analyses, including the NOAK study on the adult side, have shown a significantly better effect on asthma exacerbations with FeNO-guided treatment, in both children and adults [13]. However, our study is the only one thus far performed within primary care. Furthermore, in a post hoc analysis of the NOAK study, we could also show that the levels of total IgE and IgE antibodies against, for example, furred pets, decreased over the course of 12 months with optimised treatment [14]. The decrease of IgE correlated with decrease of FeNO, and with improved asthma control and asthma-related quality of life.

As indicated above, FeNO may provide important information to the physician about the patient's treatment adherence and possible effects of allergen exposure. Further, reporting the FeNO value to the patient may increase the patient's awareness about his/her disease, possibly leading to change in behaviour. These are aspects of FeNO measurements that cannot be captured in a randomized, controlled trial such as the NOAK study described above. Therefore, we are now planning for a real-world cluster-randomized, controlled study within primary health care, to be able to catch also these aspects of FeNO measurements. Only one previous study has aimed at such study design [15]. However, due to the lack of FeNO-naïve allergy clinics in the area, true cluster-randomization could not be done, leading to baseline bias, and the study was partly negative. In Stockholm County, this will not constitute a problem since no single primary health care center use FeNO measurements today in this region.

Aim The overall aim of this real-world, cluster-randomised study is to investigate if use of FeNO measurements in primary care, to guide anti-inflammatory treatment, can improve treatment outcome and care of adult patients with asthma.

Research questions All research questions relate to use of FeNO measurements in primary care for monitoring of anti-inflammatory treatment in individuals aged ≥ 18 years with asthma/suspected asthma.

Primary research question

- Can use of FeNO measurements decrease the number of exacerbations?

Secondary research questions

* Can use of FeNO measurements improve asthma control as measured using the Asthma Control Test (ACT) questionnaire?
* Can use of FeNO measurements improve lung function, measured using spirometry, as regards FEV1 (forced expiratory volume in one second) and FEV1 in percent of expected (reference values from Hedenström)?
* Can use of FeNO measurements decrease the use of short-acting β2 receptor agonists (salbutamol, terbutaline and formoterol)?
* Can use of FeNO measurements decrease the total cost of drugs for asthma treatment?

The study could lead to more certain asthma diagnoses, better treatment adherence and more optimised anti-inflammatory treatment. If the study can indicate positive effects for patients with asthma in regular clinical practice in primary care, the results may lead to changed national recommendations on asthma patient care (Swedish National Board of Health and Wellfare).

Work plan Study design: The study is devised as a real-world cluster randomised intervention study. Healthcare centres within Stockholm County with at least 7,000 listed patients, which use the medical record system TakeCare and have a certified asthma/COPD facility, can participate in the study. Eligible Healthcare centres should also on a routine basis transfer data to the Swedish National Airway Register. The power calculation for the study in this application is based on the NOAK study, with exacerbation frequency as the primary outcome measure. In a trial with 6 clusters per arm, the total minimum sample size was determined to be 636 (on average 53 patients per cluster), to obtain 80% power (alpha=0.05), and to detect a 10 per cent unit reduction in exacerbation rate. The participating healthcare centres will be randomised to two equal-sized groups, one intervention group and one control group, and will be followed for two years.

Intervention: Physicians, nurses and other staff at the healthcare centres in the intervention group will get a two-hour education on what FeNO is, how a FeNO measurement is performed, and how FeNO values can be interpreted and used to guide anti-inflammatory treatment. A web-based FeNO Interpretation Aid to assist in determining if a value is elevated or not, with individual tailoring based on gender, age and height, will be provided. We have previously shown that reference equations can be developed using Lambda-Mu-Sigma models, similar to Global Lung Function Initiative [16]. In The FeNO Interpretation Aid we will use data from both the US (NHANES) and Sweden. A follow-up meeting, approximately one hour in length, is planned for one month after the education, to enable evaluation and provide the opportunity to ask questions. The healthcare centres in the control group will continue to care for their asthma patients as usual.

For the patients in the intervention group, the study means that they will have to perform a FeNO measurement for the asthma/COPD nurse in connection with an asthma-related visit to the healthcare centre, when this is considered justified. A FeNO measurement involves a maximal inhalation, followed by an even exhalation for ten seconds into a FeNO measuring device. The results are shown on a display after about one minute. The asthma/COPD nurse enters the result of a FeNO measurement into the patient's medical record. The treating physician can then assess the result and decide on any change to the anti-inflammatory treatment.

Data collection: Approval from the ethics board and written approval from each centre's manager are required. The asthma/COPD nurses extract medical record data after one and two years, in accordance with items 1-6 below, from the healthcare centres' medical record system TakeCare using the data collection program MedRave4. The data collected are exported to Excel on the asthma/COPD nurses' computers and all personal data are erased.

1. Number of patients aged ≥ 18 years, with a diagnosis of asthma in the past year, plus their gender and age.
2. Number of recorded exacerbation diagnoses.
3. Points on the Asthma Control Test questionnaire.
4. Spirometry results (FEV1 in litres and in percent of expected value).
5. Results of FeNO measurements performed (active centers).

Data on filled prescriptions, to calculate drug use and costs, will be collected at the healthcare centre level through the follow-up portal GUPS, which can be accessed online through the portal Janusinfo (www.janusinfo.se) under drug statistics. With the approval of the GUPS system owner and the healthcare centre's manager, data for each individual healthcare centre can be collected. These data can be connected to diagnosis using the so-called VAL database, for which we can get assistance from the Drug and Therapeutics Committee in Region Stockholm. From the Swedish National Airway Register the following variables will be collected: Date of examination, Sex, Age, Asthma diagnosis (year), Allergy diagnosis (year), Height, Weight, Body Mass Index, Smoke habits, Spirometry measures, Number of asthma exacerbations last 12 months, Number of hospitalizations because of asthma last 12 months, Received patient asthma education, Asthma Control Test score, Asthma severity, FeNO value, Objective allergy testing (year), Respiratory allergy, Asthma or Allergy medication categories and Other Allergy manifestations. Descriptive data on the healthcare centres, such as the number of listed patients, operative form, asthma/COPD facilities, further education, and socio-demographics, are collected through interviews with the asthma/COPD nurses. After this, analyses and statistical processing can be performed.

References

1. Miljöhälsorapport 2013. , in Institutet för miljömedicin KI. 2013. p. ki.se/sites/default/files/mhr2013.pdf.
2. Nathan RA, Meltzer EO, Blaiss MS, Murphy KR, Doherty DE, and Stoloff SW, Comparison of the Asthma in America and Asthma Insight and Management surveys: did asthma burden and care improve in the United States between 1998 and 2009? Allergy Asthma Proc, 2012. 33 (1): 65-76.
3. Stallberg B, Lisspers K, Hasselgren M, Janson C, Johansson G, and Svardsudd K, Asthma control in primary care in Sweden: a comparison between 2001 and 2005. Prim Care Respir J, 2009. 18 (4): 279-86.
4. Alving K, Weitzberg E, and Lundberg JM, Increased amount of nitric oxide in exhaled air of asthmatics. Eur Respir J, 1993. 6 (9): 1368-70.
5. Malinovschi A, Fonseca JA, Jacinto T, Alving K, and Janson C, Exhaled nitric oxide levels and blood eosinophil counts independently associate with wheeze and asthma events in National Health and Nutrition Examination Survey subjects. J Allergy Clin Immunol, 2013. 132 (4): 821-827 e5.
6. Pavord ID and Bafadhel M, Exhaled nitric oxide and blood eosinophilia: independent markers of preventable risk. J Allergy Clin Immunol, 2013. 132 (4): 828-9.
7. Asthma: diagnosis, monitoring and chronic asthma management. NICE Guidance (British National Institute for Health and Care Excellence), 2016: https://www.nice.org.uk/guidance/ng80.
8. Sverrild A, Malinovschi A, Porsbjerg C, Backer V, and Alving K, Predicting airway hyperreactivity to mannitol using exhaled nitric oxide in an unselected sample of adolescents and young adults. Respir Med, 2013. 107 (1): 150-2.
9. Price DB, Buhl R, Chan A, Freeman D, Gardener E, Godley C, Gruffydd-Jones K, McGarvey L, Ohta K, Ryan D, Syk J, Tan NC, Tan T, Thomas M, Yang S, Konduru PR, Ngantcha M, d'Alcontres MS, and Lapperre TS, Fractional exhaled nitric oxide as a predictor of response to inhaled corticosteroids in patients with non-specific respiratory symptoms and insignificant bronchodilator reversibility: a randomised controlled trial. Lancet Respir Med, 2018. 6 (1): 29-39.
10. Nolte H, Pavord I, Backer V, Spector S, Shekar T, Gates D, Nair P, and Hargreave F, Dose-dependent anti-inflammatory effect of inhaled mometasone furoate/formoterol in subjects with asthma. Respir Med, 2013. 107 (5): 656-64.
11. Syk J, Unden AL, and Alving K, Relationship between exhaled nitric oxide and IgE sensitisation in patients with asthma: influence of steroid treatment. Clin Respir J, 2009. 3 (3): 143-51.
12. Syk J, Malinovschi A, Johansson G, Unden AL, Andreasson A, Lekander M, and Alving K, Anti-inflammatory treatment of atopic asthma guided by exhaled nitric oxide: a randomized, controlled trial. J Allergy Clin Immunol Pract, 2013. 1 (6): 639-48 e1-8.
13. Petsky HL, Cates CJ, Kew KM, and Chang AB, Tailoring asthma treatment on eosinophilic markers (exhaled nitric oxide or sputum eosinophils): a systematic review and meta-analysis. Thorax, 2018. 73 (12): 1110-1119.
14. Syk J, Malinovschi A, Borres MP, Unden AL, Andreasson A, Lekander M, and Alving K, Parallel reductions of IgE and exhaled nitric oxide after optimized anti-inflammatory asthma treatment. Immun Inflamm Dis, 2016. 4 (2): 182-190.
15. Zeiger RS, Schatz M, Yang SJ, and Chen W, Fractional Exhaled Nitric Oxide-Assisted Management of Uncontrolled Persistent Asthma: A Real-World Prospective Observational Study. Perm J, 2019. 23.
16. Jacinto T, Amaral R, Malinovschi A, Janson C, Fonseca J, and Alving K, Exhaled NO reference limits in a large population-based sample using the Lambda-Mu-Sigma method. J Appl Physiol (1985), 2018. 125 (5): 1620-1626.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma according to medical record.
* Patients seeking advice for symptoms suggestive of asthma

Exclusion Criteria:

* Physician diagnosed COPD (Chronic Obstructive Pulmonary Disease) according to medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Exacerbation rate | Two years
  Can use of FeNO measurements decrease the number of exacerbations compared to usual care.

SECONDARY OUTCOMES:
Asthma control | Two years
  Can use of FeNO measurements improve asthma control as measured using the Asthma Control Test (ACT) questionnaire, compared to usual care.
Lung function | Two years
  Can use of FeNO measurements improve lung function, measured using spirometry, as regards FEV1 (forced expiratory volume in one second) and FEV1 in percent of expected (reference values from Hedenström), compared to usual care.
Use of short-acting β2 receptor agonists | Two years
  Can use of FeNO measurements decrease the use of short-acting β2 receptor agonists (salbutamol, terbutaline and formoterol), compared to usual care.
Total cost of asthma medications | Two years
  Can use of FeNO measurements decrease the total cost of drugs for asthma treatment, compared to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Jörgen Syk, MD PhD, Principal Investigator — Region Stockholm
Locations (1):
- Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No